CLINICAL TRIAL: NCT07300618
Title: The Effect of Stress Ball And Music on Anxiety, Stress, and Pain Levels During Platelet Apheresis Donation: Randomized Controlled Trial
Brief Title: Stress Ball and Music to Reduce Anxiety and Pain in Platelet Apheresis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Dilek Urtekin, PhD, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023.03.01.03
Record Dates: First submitted 2025-11-17; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Anxiety; Stress
Keywords: Platelet apheresis; Anxiety; Stress; Nursing
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- müzik resital (Experimental): During the platelet apheresis donation, instrumental music was played for the participant for 30 minutes.
  Interventions: Other: müzik resital; Device: aferez makinesi; Drug: antikoagülan çözelti
- stres topu (Experimental): The participant was instructed to squeeze a stress ball for 30 minutes during the platelet apheresis donation.
  Interventions: Other: stres topu; Device: aferez makinesi; Drug: antikoagülan çözelti
- kontrol grubu (No Intervention): Routine treatment and follow-up were continued, and no intervention was applied.

INTERVENTIONS:
Other: müzik resital — After the platelet apheresis procedure began, donors in the music listening group were exposed to instrumental music composed of Classical Turkish Music modes for 30 minutes through the center's speaker system.
  Arms: müzik resital
Other: stres topu — When the platelet apheresis procedure began, a stress ball was placed in the palm of one hand of the donors in the stress ball group. They were instructed to squeeze the ball at their preferred frequency for a total of 30 minutes during the apheresis procedure.
  Arms: stres topu
Device: aferez makinesi — The platelet apheresis procedure was performed on donors using an apheresis machine.
  Other Names: Spektral Optik
  Arms: müzik resital; stres topu
Drug: antikoagülan çözelti — In accordance with the operating principle of the platelet apheresis device, the anticoagulant solution ACD-A is routinely used for all donors.
  Other Names: ACD-A
  Arms: müzik resital; stres topu

SUMMARY:
This study was conducted as a single-center, prospective, randomized controlled trial to investigate the effects of stress ball use-a distraction and attention-directing method-and music listening, which targets the auditory sensory pathway, on anxiety, stress, and pain levels in platelet apheresis donors beyond routine care. The study sample consisted of 102 donors aged 18 to 55 years who were donating platelets for the first time at a university hospital blood transfusion center. The participants were divided into three groups: 34 in the stress ball group, 34 in the music listening group, and 34 in the control group. Data were collected using the Donor Information Form, the Beck Anxiety Inventory (BAI), the Visual Analogue Scale (VAS) for pain, the Distress Thermometer (DT), and the Donor Follow-up Chart. During platelet apheresis, participants in the stress ball group were instructed to squeeze a stress ball for 30 minutes, those in the music group listened to instrumental music for 30 minutes, and the control group received only routine care without any additional intervention.

DETAILED DESCRIPTION:
Data Collection and Evaluation Process Pre-Implementation Phase Before starting the study, a pilot test was conducted with 10% of the individuals representing the study sample to evaluate the understandability and usability of the scales and forms to be used as data collection tools, as well as to assess the feasibility of stress ball and music interventions. Based on the results of the pilot study, necessary revisions were made to the study content, forms, stress ball application, and music intervention, and the final version of the study protocol was created. Data obtained from the pilot study were not included in the main analysis. Implementation Phase Donors who met the inclusion criteria were informed by the researchers about the purpose, design, and method of the study. Written informed consent was obtained from all participants using separate Informed Consent Forms prepared for each group. Stress Ball Group Ten minutes before the platelet apheresis procedure, participants completed the Donor Information Form, Beck Anxiety Inventory (BAI), Distress Thermometer (DT), and Visual Analog Scale (VAS) as a pre-test through face-to-face interviews. Vital signs were recorded on the Donor Monitoring Chart. When the platelet apheresis procedure began, a stress ball was placed in the donor's hand. Participants were instructed to squeeze the ball at their preferred frequency for a total of 30 minutes during the apheresis procedure. Five minutes after the donation was completed, the BAI, DT, and VAS were administered again as post-tests. Vital signs were recorded on the Donor Follow-up Table, indicating that the study procedure was complete.

Music Listening Group Ten minutes before the platelet apheresis procedure, participants completed the Donor Information Form, Beck Anxiety Inventory (BAI), Distress Thermometer (DT), and Visual Analogue Scale (VAS) as pre-tests through face-to-face interviews. Their vital signs were recorded on the Donor Follow-up Chart. After the platelet apheresis procedure began, instrumental music composed of Classical Turkish Music modes was played for 30 minutes through the center's speaker system. Five minutes after the donation was completed, the BAI, DT, and VAS were administered again as post-tests. Vital signs were recorded, and the study procedure was concluded.

Control Group Ten minutes before the platelet apheresis procedure, participants completed the Donor Information Form, BAI, DT, and VAS as pre-tests through face-to-face interviews. Their vital signs were recorded on the Donor Follow-up Chart. During the platelet apheresis procedure, no additional intervention was applied to the donors in the control group, and they continued to receive routine care. Five minutes after the procedure was completed, the BAI, DT, and VAS were administered again as post-tests. Vital signs were recorded, and the study was concluded.

Ethical Considerations Ethical approval for the study was obtained from the institutional ethics committee (research protocol number: 2023.03.01.03). Written permission was also obtained from the institution where the study was conducted. The identities of the researchers and the data obtained from the study were kept confidential.

ELIGIBILITY:
Inclusion Criteria

Donors who:

* Were literate in Turkish
* Had no physical limitations preventing them from squeezing a stress ball
* Had no psychiatric disorders or visual, auditory, or perceptual impairments
* Met the institution's platelet apheresis donation criteria
* Were donating platelets for the first time
* Voluntarily wished to donate platelets
* Agreed to participate in the study

Exclusion Criteria

Donors who:

* Withdrew from platelet apheresis donation
* Wished to withdraw from the study
* Developed a reaction during the donation
* Had insufficient blood flow through the catheter
* Were unable to complete the platelet apheresis donation

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-11-20 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Pain Intensity Measured by the Visual Analogue Scale (VAS) | 30 minutes
  The Visual Analogue Scale (VAS) is a validated, self-reported measure used to assess pain intensity. The scale ranges from 0 to 10, where 0 indicates no pain and 10 indicates the worst possible pain. Higher scores represent greater pain intensity. Pain will be measured immediately before and immediately after the platelet apheresis procedure.
Anxiety Levels Measured by the Beck Anxiety Inventory (BAI) | 30 minutes
  The Beck Anxiety Inventory (BAI) is a 21-item, self-reported questionnaire used to assess the severity of anxiety symptoms. Each item is scored from 0 to 3, producing a total score ranging from 0 to 63. Higher scores indicate higher levels of anxiety. Anxiety will be measured immediately before and immediately after the platelet apheresis procedure in all groups.
Stress Levels Measured by the Distress Thermometer (DT) | 30 minutes
  The Distress Thermometer (DT) is a validated, self-reported screening tool used to assess stress and distress levels. It consists of a single-item visual scale ranging from 0 to 10, where 0 indicates no stress/distress and 10 indicates extreme stress/distress. Higher scores represent higher levels of stress. Stress levels will be measured immediately before and immediately after the platelet apheresis procedure in all groups.

CONTACTS AND LOCATIONS:
Overall Officials: Seval SA Akpınar, Seval a, Study Director — namık kemal üniversitesi
Locations (1):
- Tekirdağ Namık Kemal University, Tekirdağ, Süleymanpaşa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I prefer not to

REFERENCES:
- [Background] Wen X, Shi J, Tan W, Jiang H, Wang D, Su J, Yang G, Zhang B. Effects of aromatherapy and music therapy on patients' anxiety during MRI examinations: a randomized controlled trial. Eur Radiol. 2023 Apr;33(4):2510-2518. doi: 10.1007/s00330-022-09230-3. Epub 2022 Nov 6. PMID 36335480
- [Background] Abdul Hamid MR, Mansor MB, Zainal Abidin MF. Music therapy for reducing anxiety in patients undergoing total knee replacement surgery under subarachnoid anesthesia. J Orthop Surg (Hong Kong). 2022 May-Aug;30(2):10225536221122347. doi: 10.1177/10225536221122347. PMID 36031855
- [Background] Yanes AF, Weil A, Furlan KC, Poon E, Alam M. Effect of Stress Ball Use or Hand-holding on Anxiety During Skin Cancer Excision: A Randomized Clinical Trial. JAMA Dermatol. 2018 Sep 1;154(9):1045-1049. doi: 10.1001/jamadermatol.2018.1783. PMID 30027283
- [Background] Duncanson E, Le Leu RK, Shanahan L, Macauley L, Bennett PN, Weichula R, McDonald S, Burke ALJ, Collins KL, Chur-Hansen A, Jesudason S. The prevalence and evidence-based management of needle fear in adults with chronic disease: A scoping review. PLoS One. 2021 Jun 10;16(6):e0253048. doi: 10.1371/journal.pone.0253048. eCollection 2021. PMID 34111207
- [Background] Kabacoff RI, Segal DL, Hersen M, Van Hasselt VB. Psychometric properties and diagnostic utility of the Beck Anxiety Inventory and the State-Trait Anxiety Inventory with older adult psychiatric outpatients. J Anxiety Disord. 1997 Jan-Feb;11(1):33-47. doi: 10.1016/s0887-6185(96)00033-3. PMID 9131880
- [Background] Gezginci E, Iyigun E, Kibar Y, Bedir S. Three Distraction Methods for Pain Reduction During Cystoscopy: A Randomized Controlled Trial Evaluating the Effects on Pain, Anxiety, and Satisfaction. J Endourol. 2018 Nov;32(11):1078-1084. doi: 10.1089/end.2018.0491. PMID 30280915
- [Background] Cline ME, Herman J, Shaw ER, Morton RD. Standardization of the visual analogue scale. Nurs Res. 1992 Nov-Dec;41(6):378-80. No abstract available. PMID 1437591

DOCUMENTS (4):
  • Study Protocol and Statistical Analysis Plan (2023-01-31): https://cdn.clinicaltrials.gov/large-docs/18/NCT07300618/Prot_SAP_000.pdf
  • Informed Consent Form: Control Group (2023-01-31): https://cdn.clinicaltrials.gov/large-docs/18/NCT07300618/ICF_001.pdf
  • Informed Consent Form: Music Resital Group (2023-01-31): https://cdn.clinicaltrials.gov/large-docs/18/NCT07300618/ICF_002.pdf
  • Informed Consent Form: Stress Ball Group (2023-01-31): https://cdn.clinicaltrials.gov/large-docs/18/NCT07300618/ICF_003.pdf